CLINICAL TRIAL: NCT04150029
Title: A Phase II Multi-center, Single Arm, Safety and Efficacy Study of MBG453 in Combination With Azacitidine and Venetoclax for the Treatment of Acute Myeloid Leukemia (AML) in Adult Patients Unfit for Chemotherapy
Brief Title: A Study of MBG453 in Combination With Azacitidine and Venetoclax in AML Patients Unfit for Chemotherapy
Acronym: STIMULUS-AML1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Novartis made a decision to early terminate the sabatolimab clinical development program, including the CMBG453C12201 trial, following the negative results from other 2 trials.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453C12201; 2019-000439-14 (EudraCT Number)
Record Dates: First submitted 2019-10-22; First posted 2019-11-04 (Actual); Results first posted 2025-11-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: MBG453; Venetoclax; Azacitidine; Phase 2; AML; Acute myeloid Leukemia; Sabatolimab
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — sabatolimab; venetoclax; Azacitidine

STUDY DESIGN:
Intervention Model Description: safety -run -in with escalating dose of MBG453 followed by expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MBG453+Venetoclax +Azacitidine (Experimental): Participants received MBG453 in combination with Venetoclax and Azacitidine
  Interventions: Drug: MBG453; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: MBG453 — Solution for intravenous infusion
  Other Names: Sabatolimab
Drug: Venetoclax — Tablet for oral administration
Drug: Azacitidine — Solution for subcutaneous injection or intravenous infusion

SUMMARY:
This trial seeked to extend the preliminary findings of efficacy by evaluating MBG453 in combination with hypomethylating agents (HMA) and also Bcl-2 inhibitor venetoclax.

DETAILED DESCRIPTION:
The primary purpose of Part 1 (Safety Run-in) was to rule out excessive toxicity of MBG453, when administered in combination with azacitidine and venetoclax.

The primary purpose of the combined Part 1 and Part 2 (Safety run-in and Expansion Part) was to evaluate efficacy of MBG453, when administered in combination with azacitidine and venetoclax in adult patients with newly diagnosed AML, who were not suitable for treatment with intensive chemotherapy.

Originally, there was an analysis planned of the complete response (CR) rate, after all subjects had completed at least 12 cycles of treatment (each cycle = 28 Days) or discontinued earlier. As Novartis decided to end the development of this compound, this primary analysis was skipped and only the final study analysis presented here. At the final analysis timepoint, there was only 1 patient who didn't completed the 12 cycles of treatment or discontinued earlier.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Age ≥ 18 years at the date of signing the informed consent form (ICF)
* Newly diagnosed with AML based on 2016 WHO classification (Arber et al 2016) and not suitable for intensive chemotherapy defined as: age ≥75, ECOG performance Status 2 or 3, or any of the following comomorbitities: severe cardiac comorbities (including congestive heart failure, LVEF ≤ 50%, chronic stable Angina) , pulmonary comorbidity (DLCO ≤ 65% or FEVI ≤ 65%). moderate hepatic impairment (with total Bilirubin >1.5 to 3x ULN) , renal impairment (eGFR≥ 30 ml/min/1.73m^2 to <45 ml/min/1.73m^2), or other comorbidity incompatible with intensive chemotherapy per Investigator assessement and approved by the Novartis Medical monitor)
* Not planned for hematopoietic stem-cell transplantation (HSCT)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 , 2 or 3

Exclusion Criteria:

* Prior exposure to TIM-3 directed therapy
* History of severe hypersensitivity reactions to any ingredient of study drug(s) (azacitidine, venetoclax or MGB453) or monoclonal antibodies (mAbs) and/or their excipients
* Current use or use within 14 days prior to randomization of systemic, steroid therapy (> 10 mg/day prednisone or equivalent) or any immunosuppressive therapy. Topical, inhaled, nasal, ophthalmic steroids are allowed. Replacement therapy, steroids given in the context of a transfusion are allowed and not considered a form of systemic treatment.
* Previous treatment at any time, with any of the following antineoplastic agents, approved or investigational; checkpoint inhibitors, venetoclax and hypomethylating agents (HMAs) such as decitabine or azacitidine.
* Active autoimmune disease requiring systemic therapy (e.g.corticosteroids).
* Live vaccine administered within 30 Days prior to randomization

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (28):
- United States (12):
  - 25Uni of Alabama at Birmingham, Birmingham, Alabama
  - Yale University School Of Medicine, New Haven, Connecticut
  - Uni Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering, New York, New York
  - Weill Cornell Medicine NY-Presb, New York, New York
  - Levine Cancer Insitute Carolinas Healthcare System, Charlotte, North Carolina
  - Duke Univ Medical Center, Durham, North Carolina
  - Chattanooga Onc And Hem Assoc PC, Chattanooga, Tennessee
  - MD Anderson Cancer Center University of Texas, Houston, Texas
  - Huntsman Cancer Institute Univ of Utah, Salt Lake City, Utah
- Novartis Investigative Site, Clayton, Victoria, Australia
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Berlin
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
- Japan (2):
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Yamagata, Yamagata
- Novartis Investigative Site, Seoul, Seocho gu, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 28 centers across 10 countries with a total of 90 participants enrolled.
Pre-assignment Details: Informed consent was obtained from each participant in writing before screening before any study specific procedure was performed.
Groups:
- MBG453 400 mg + Venetoclax +Azacitidine: Participants received 400 mg MBG453 in combination with Venetoclax (VEN) and Azacitidine (AZA). This arm was used in Part 1 (Safety Run-in phase) of the study.
- MBG453 800 mg + Venetoclax +Azacitidine: Participants received 800 mg MBG453 in combination with Venetoclax (VEN) and Azacitidine (AZA). This arm was used in Part 1 (Safety Run-in phase) and Part 2 (Expansion Part) of the study.
Period: Overall Study
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Started | 5 | 85
Did not enter post-treatment follow-up | 4 | 60
Entered post-treatment follow-up | 1 | 25
Entered survival follow-up | 5 | 85
Completed (Completed = completed treatment) | 0 | 0
Not Completed | 5 | 85
Not completed — Disease Relapse | 0 | 18
Not completed — Progressive Disease | 2 | 16
Not completed — Adverse Event | 1 | 11
Not completed — Physician Decision | 0 | 10
Not completed — Study Terminated by Sponsor | 1 | 10
Not completed — Death | 0 | 8
Not completed — Participant Decision | 0 | 7
Not completed — Hemopoietic Stem Cell Transplant (HSCT) | 1 | 5

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax).
Groups:
- Total: Total of all reporting groups
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine | Total
Number analyzed (Participants) | 5 | 85 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.8 (4.97) | 76.1 (6.33) | 76.1 (6.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 38 | 39
  Male | 4 | 47 | 51
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 69 | 74
  Black or African American | 0 | 2 | 2
  Asian | 0 | 13 | 13
  Unknown | 0 | 1 | 1
Body surface area (BSA) [Mean (Standard Deviation); unit: m^2] — BSA is a measurement of the total area of the skin of a human body, usually expressed in square meters (m²). It's a crucial parameter in various medical calculations, including drug dosages, fluid administration, and determining metabolic mass. BSA (m^2) at baseline is calculated as square root of (weight (kg) * height (cm)/3600) using weight at baseline and height at screening.
  m^2 | 1.88 (0.105) | 1.84 (0.252) | 1.84 (0.246)
ECOG performance status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status scale is a widely used standard of care criteria used to assess the functional status of a patient with cancer to measure how the disease impacts thepatient's daily living abilities. This scale has a range from 0 - 5. The higher the grade, the worse the patient's abilities: 0 implies fully active, able to carry on all pre-disease performance without restriction and 5 implies death.
  Participants
    ECOG performance status: 0 | 1 | 14 | 15
    ECOG performance status: 1 | 2 | 43 | 45
    ECOG performance status: 2 | 2 | 24 | 26
    ECOG performance status: 3 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Dose Limiting Toxicities (DLT)(Safety run-in Patients Only)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value considered by the Investigator to be at least possibily related to MBG453 as a single contributor or in combination with other component(s) of study treatment that occurs during the DLT observation period and meets any of the criteria as per protolcol.
Time Frame: From Cycle 1 Day 8 to end of Cycle 2; Cycle =28 Days
Population: The Dose-Determining Set (DDS) included all participants from the FAS enrolled in the safety run-in part who met the minimum exposure criterion and had sufficient safety evaluations or experienced a dose limiting toxicity (DLT) starting from Cycle 1 Day 8 to the end of Cycle 2.
  FAS comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax).
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 4 | 11
Participants
  Participants with at least 1 event - All grades | 0 | 1
  Participants with at least 1 event - Grade >= 3 | 0 | 0
  Cardiac disorders - All grades | 0 | 1
  Cardiac disorders - Grades >= 3 | 0 | 0

2. Primary Outcome: Percentage of Participants Achieving Complete Remission (CR) (CR Rate)
Description: CR rate is defined as the percentage of participants achieving a complete remission (CR) as per investigator assessment (based on IWG Cheson et al 2003, ELN 2017 Dohner et al 2017).
Time Frame: approx. 31 months
Population: All participants in the Full Analysis Set (FAS) and assigned to MBG453 at the 800 mg Q4W dose level. FAS comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 85
Percentage of participants | 47.06 [36.1 to 58.2]

3. Secondary Outcome: Measurable Residual Disease (MRD) - Negativity Rate: Full Study Population
Description: MRD negativity rate was defined as the percentage of participants with MRD negativity, which was defined as an MRD negative sample (frequency of LAIP below 0.1%, as determined by Multi-parameter Flow Cytometry-Measurable residual disease (MFC-MRD) at Central Lab) in participant with remission (i.e., CR or CRi) as per investigator assessment (based on IWG Cheson et al 2003, ELN 2017 Dohner et al 2017). MRD-negative response was required to be observed at or after morphological remission, and prior to relapse or disease progression.
Time Frame: approx. 31 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Percentage of participants | 60.0 [14.7 to 94.7] | 42.4 [31.7 to 53.6]

4. Secondary Outcome: Measurable Residual Disease (MRD) - Negativity Rate in Participants With Best Overall Response (BOR) of CR/CRi and Evaluable MRD
Description: as for outcome 3
Time Frame: approx. 31 months
Population: All participants in FAS with the best overall response of CR or CRi and who are evaluable for MRD. The Full Analysis Set (FAS) comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax). A participant is considered as evaluable for MRD if he/she had at least one post-baseline sample with MRD negative or MRD positive.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 3 | 49
Percentage of participants | 100.0 [29.2 to 100.0] | 73.5 [58.9 to 85.1]

5. Secondary Outcome: Duration of Complete Remission (CR)
Description: The duration of CR is defined as the time from first achievement of CR to the first documented relapse or progressive disease or death due to any cause, whichever occurs first. The response assessment is as per investigator assessment based on IWG (Cheson et al 2003) and ELN 2017 (Dohner et al 2017).
Time Frame: approx. 31 months
Population: The Full Analysis Set (FAS) comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax). This was based on participants with best overall response of CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 4 | 40
Months | NA [7.56 to NA] — NA: median and upper limit of confidence interval was not achieved due to small sample size and short duration of follow-up. | 10.28 [6.28 to NA] — NA: upper limit of confidence interval was not achieved due to small sample size and short duration of follow-up.

6. Secondary Outcome: Percentage of Participants Achieving a Complete Remission (CR) or Complete Remission With Incomplete Hematologic Blood Count Recovery (CRi) (CR/CRi Rate)
Description: CR/CRi rate is defined as the percentage pf participants with best overall response of either complete remission (CR) or complete remission with incomplete hematologic recovery (CRi) as per investigator assessment (based on IWG (Cheson et al 2003) and ELN 2017 (Dohner et al 2017)).
Time Frame: approx. 31 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Percentage of participants | 80.0 [28.4 to 99.5] | 69.4 [58.5 to 79.0]

7. Secondary Outcome: The Duration of Complete Remission (CR)/Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: The duration of CR/CRi is defined as the time from first achievement of CR or CRi to the first documented relapse or progressive disease or death due to any cause, whichever occurs first. The response assessment is as per investigator assessment based on IWG (Cheson et al 2003) and ELN 2017 (Dohner et al 2017).
Time Frame: approx. 31 months
Population: The Full Analysis Set (FAS) comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax). This was based on participants with best overall response of CR or CRi.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 4 | 59
Months | NA [7.56 to NA] — NA: Median and upper limit of CI were not achieved due to small sample size and short duration of follow-up. | 8.54 [5.98 to 13.67]

8. Secondary Outcome: Percentage of Participants Achieving a Complete Remission (CR) or Complete Remission With Partial Hematologic Blood Count Recovery (CRh) (CR/CRh Rate)
Description: CR/CRh rate is defined as the percentage of participants with best overall response of either complete remission (CR) or complete remission with partial hematologic recovery (CRh) as per derivation based on ELN 2022 (Döhner et al 2022).
Time Frame: approx. 31 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Percentage of participants | 80.0 [28.4 to 99.5] | 50.6 [39.5 to 61.6]

9. Secondary Outcome: Duration of CR/CRh
Description: The duration of CR/CRh is defined as the time from date of first documented CR or CRh to the date of first documented relapse or death due to any cause, whichever occurs first. The response assessment is as per derivation based on ELN 2022 (Döhner et al 2022).
Time Frame: approx. 31 months
Population: The Full Analysis Set (FAS) comprised all participants who received at least one dose of any component of the study treatment (i.e. at least one dose of sabatolimab or at least one dose of azacitidine or at least one dose of venetoclax). This was based on participants with best overall response of CR or CRh.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 4 | 43
Months | NA [7.56 to NA] — NA: Median and upper limit of confidence interval were not achieved due to small sample size and short duration of follow-up. | 12.45 [6.83 to 14.78]

10. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is the time from start of treatment until death due to any cause, relapse from complete remission (CR) or complete remission with incomplete hematologic recovery (CRi), or treatment failure, whichever occurs first. Treatment failure was defined as lack of reaching CR until Cycle 8 Day 1 or earlier permanent discontinuation from study without reaching CR, the time to treatment failure was then set to Day 1.
Time Frame: approx. 31 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Months | 8.28 [0.03 to NA] — NA: upper limit of confidence interval was not achieved due to small sample size and short duration of follow-up. | 0.03 [0.03 to 6.14]

11. Secondary Outcome: Overall Survival (OS)
Description: OS is the time from start of treatment to death due to any cause. If a participant was not known to have died, then OS was censored at the latest date the participant was known to be alive (on or before the cut-off date).
Time Frame: approx. 31 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Months | 11.17 [5.32 to NA] — NA: Upper limit of confidence interval was not achieved due to small sample size and short duration of follow-up. | 13.27 [9.49 to 18.14]

12. Secondary Outcome: Peak Serum Concentration (Cmax) of MBG453
Description: Cmax is the maximal concentration of MBG453.
Time Frame: Cycle 1 Day 8 (end of infusion) and Cycle 3 Day 8 (end of infusion), cycle = 28 days
Population: The sabatolimab pharmacokinetic analysis set included all participants from the Safety Set who provided at least one evaluable sabatolimab PK concentration for the two populations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 81
ug/ml
  Cycle 1 Day 8: 2 hr (post-dose): number analyzed (Participants) | 4 | 67
  Cycle 1 Day 8: 2 hr (post-dose) | 84.0 (20.0) | 204 (35.3)
  Cycle 3 Day 8: 2 hr (post-dose): number analyzed (Participants) | 2 | 46
  Cycle 3 Day 8: 2 hr (post-dose) | 129 (4.9) | 261 (40.9)

13. Secondary Outcome: Trough Serum Concentration (Cmin) MBG453
Description: Cmin is the minimum concentration of MBG453 (i.e., prior to the next dosing).
Time Frame: Day 8 of Cycle 1,2,3,6,9,12,18, 24 and through treatment completion, an average of 24 months
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/ml
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 81
ug/ml
  Cycle 1 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 5 | 73
  Cycle 1 Day 8: 0 hr (pre-dose) | 0 (0) | 0 (0)
  Cycle 2 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 4 | 61
  Cycle 2 Day 8: 0 hr (pre-dose) | 8.79 (70.8) | 18.8 (68.9)
  Cycle 3 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 2 | 51
  Cycle 3 Day 8: 0 hr (pre-dose) | 12.4 (16.0) | 30.7 (80.9)
  Cycle 6 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 2 | 26
  Cycle 6 Day 8: 0 hr (pre-dose) | 17.6 (0) | 45.1 (79.5)
  Cycle 9 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 1 | 17
  Cycle 9 Day 8: 0 hr (pre-dose) | 6.55 (0) | 72.9 (60.0)
  Cycle 12 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 1 | 10
  Cycle 12 Day 8: 0 hr (pre-dose) | 17.4 (0) | 78.1 (62.7)
  Cycle 18 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 1 | 7
  Cycle 18 Day 8: 0 hr (pre-dose) | 9.76 (0) | 70.4 (96.5)
  Cycle 24 Day 8: 0 hr (pre-dose): number analyzed (Participants) | 1 | 2
  Cycle 24 Day 8: 0 hr (pre-dose) | 30.6 (0) | 61.4 (84.1)

14. Secondary Outcome: Trough Plasma Concentration (Cmin) Venetoclax
Description: Trough concentration of venetoclax on treatment
Time Frame: 0 hr (Pre-dose) of Day 8 of Cycle 1, 3 and 6 ; Cycle =28 days
Population: The venetoclax pharmacokinetic analysis set included all participants from the Safety Set who provided at least one evaluable venetoclax PK concentration for the two populations.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 3 | 62
ng/ml
  Cycle 1 day 8: 0 hr pre-dose): number analyzed (Participants) | 3 | 49
  Cycle 1 day 8: 0 hr pre-dose) | 378 (86.4) | 972 (97.5)
  Cycle 3 day 8: 0 hr pre-dose): number analyzed (Participants) | 2 | 32
  Cycle 3 day 8: 0 hr pre-dose) | 730 (8.6) | 1010 (154.8)
  Cycle 6 day 8: 0 hr pre-dose): number analyzed (Participants) | 0 | 12
  Cycle 6 day 8: 0 hr pre-dose) |  | 959 (64.1)

15. Secondary Outcome: Anti-drug Antibody (ADA) Prevalence at Baseline and ADA Positive Participants On-treatment
Description: Immunogenicity (IG) to MBG453 prior to MBG453 exposure. ADA prevalence (i.e., ADA-positive samples) is the number of ADA-positive samples among the number of participants with a non-missing sample.
Time Frame: at baseline, up to 150 days after last treatment, approx. 24 months
Population: Immunogenicity Incidence Set includes all participants in the Immunogenicity prevalence set with a non-missing baseline ADA sample and at least one non-missing post-baseline ADA sample.
  The Immunogenicity prevalence set includes all participants in the Safety Set with a non-missing baseline ADA sample or at least one non-missing post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 74
Participants
  ADA prevalence at baseline (BL) | 0 | 4
  ADA-positive participants on-treatment | 1 | 9

16. Secondary Outcome: Rate of Participants Who Achieved Transfusion Independence From Baseline and While on Treatment
Description: Percentage of participants having received no RBC/Platelets transfusions during at least 8 consecutive weeks.
Time Frame: approx. 31 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Percentage of participants
  RBC: transfusion independence at post-BL | 60.0 [14.7 to 94.7] | 57.6 [46.4 to 68.3]
  Platelet transfusion independence at post-baseline | 60.0 [14.7 to 94.7] | 65.9 [54.8 to 75.8]

17. Post Hoc Outcome: All Collected Deaths
Description: Deaths were collected from treatment start until the end of the trial, approx. 31 months including post-treatment and survival follow-up period.
Time Frame: from randomization until end of trial, approx. 31 months.
Population: Clinical database population: All participants: participants who died during treatment and post-treatment.
Measure: Number; unit: Participants
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
Number analyzed (Participants) | 5 | 85
Participants
  On-treatment deaths | 1 | 11
  Post-treatment deaths: number analyzed (Participants) | 4 | 74
  Post-treatment deaths | 2 | 45
  All deaths | 3 | 56

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected from the date of first administration of study treatment to 30 days after the date of the last administration of study treatment, up to maximum duration of 42.3 months (MBG453 400mg cohort) and 37.6 months (MBG453 800mg cohort). Deaths were collected from randomization until end of trial, approx. 31 months.
Description: Any sign or symptom that occurred during the conduct of the trial and the safety follow-up. Deaths in the post-treatment survival follow-up period are not considered adverse events.
Arm/Group | MBG453 400 mg + Venetoclax +Azacitidine | MBG453 800 mg + Venetoclax +Azacitidine
All-Cause Mortality (participants affected / at risk) | 3/5 | 56/85
Serious Adverse Events (participants affected / at risk) | 4/5 | 67/85
Other Adverse Events (participants affected / at risk) | 5/5 | 85/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MBG453 400 mg + Venetoclax +Azacitidine (N=5) | MBG453 800 mg + Venetoclax +Azacitidine (N=85)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 30
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Immune-mediated pericarditis (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders and administration site conditions) | 0 | 1
Chills (General disorders and administration site conditions) | 0 | 1
General physical health deterioration (General disorders and administration site conditions) | 0 | 1
Malaise (General disorders and administration site conditions) | 0 | 1
Pyrexia (General disorders and administration site conditions) | 0 | 13
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 2
Bacteraemia (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 5
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 2
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 8
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 4
Septic shock (Infections and infestations) | 0 | 3
Splenic infection fungal (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Immune-mediated arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Vascular dementia (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MBG453 400 mg + Venetoclax +Azacitidine (N=5) | MBG453 800 mg + Venetoclax +Azacitidine (N=85)
Anaemia (Blood and lymphatic system disorders) | 2 | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 14
Neutropenia (Blood and lymphatic system disorders) | 1 | 39
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 20
Atrial fibrillation (Cardiac disorders) | 0 | 6
Tachycardia (Cardiac disorders) | 0 | 7
Abdominal pain (Gastrointestinal disorders) | 2 | 16
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 3 | 48
Diarrhoea (Gastrointestinal disorders) | 2 | 37
Dyspepsia (Gastrointestinal disorders) | 0 | 6
Haemorrhoids (Gastrointestinal disorders) | 1 | 6
Nausea (Gastrointestinal disorders) | 3 | 32
Oral pain (Gastrointestinal disorders) | 0 | 6
Proctalgia (Gastrointestinal disorders) | 0 | 6
Stomatitis (Gastrointestinal disorders) | 0 | 13
Vomiting (Gastrointestinal disorders) | 2 | 21
Asthenia (General disorders and administration site conditions) | 1 | 11
Axillary pain (General disorders and administration site conditions) | 1 | 0
Catheter site irritation (General disorders and administration site conditions) | 1 | 0
Chest discomfort (General disorders and administration site conditions) | 1 | 1
Chest pain (General disorders and administration site conditions) | 0 | 5
Chills (General disorders and administration site conditions) | 0 | 9
Fatigue (General disorders and administration site conditions) | 2 | 23
Influenza like illness (General disorders and administration site conditions) | 1 | 2
Injection site erythema (General disorders and administration site conditions) | 1 | 3
Injection site reaction (General disorders and administration site conditions) | 3 | 7
Injection site swelling (General disorders and administration site conditions) | 1 | 1
Mucosal inflammation (General disorders and administration site conditions) | 0 | 6
Oedema (General disorders and administration site conditions) | 1 | 3
Oedema peripheral (General disorders and administration site conditions) | 2 | 25
Pyrexia (General disorders and administration site conditions) | 0 | 31
COVID-19 (Infections and infestations) | 1 | 16
Cellulitis (Infections and infestations) | 0 | 5
Influenza (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 2 | 13
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 9
Contusion (Injury, poisoning and procedural complications) | 1 | 11
Fall (Injury, poisoning and procedural complications) | 0 | 8
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 6
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3
Alanine aminotransferase increased (Investigations) | 1 | 10
Aspartate aminotransferase increased (Investigations) | 1 | 7
Blood alkaline phosphatase increased (Investigations) | 1 | 5
Blood bilirubin increased (Investigations) | 0 | 9
Blood creatinine increased (Investigations) | 0 | 13
Electrocardiogram QT prolonged (Investigations) | 0 | 6
Gamma-glutamyltransferase increased (Investigations) | 1 | 8
Lipase increased (Investigations) | 0 | 5
Lymphocyte count decreased (Investigations) | 1 | 4
Neutrophil count decreased (Investigations) | 3 | 22
Platelet count decreased (Investigations) | 3 | 29
Troponin T increased (Investigations) | 0 | 6
Weight decreased (Investigations) | 1 | 14
White blood cell count decreased (Investigations) | 1 | 16
Decreased appetite (Metabolism and nutrition disorders) | 1 | 17
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 12
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 16
Dysgeusia (Nervous system disorders) | 1 | 5
Headache (Nervous system disorders) | 2 | 17
Hypoaesthesia (Nervous system disorders) | 1 | 3
Syncope (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 5
Anxiety (Psychiatric disorders) | 0 | 5
Confusional state (Psychiatric disorders) | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 9
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 12
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 6
Erythema (Skin and subcutaneous tissue disorders) | 1 | 6
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 20
Rash (Skin and subcutaneous tissue disorders) | 0 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 5
Hypertension (Vascular disorders) | 0 | 9
Hypotension (Vascular disorders) | 1 | 20
Orthostatic hypotension (Vascular disorders) | 1 | 2
Scalp haematoma (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e. data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT04150029/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT04150029/SAP_001.pdf